CLINICAL TRIAL: NCT04110106
Title: Correlation Between Quality of Life and Severity of Parkinson's Disease by Assessing an Optimal Cut-off Point on the Parkinson's Disease Questionnaire (PDQ-39) as Related to the Hoehn & Yahr (H&Y) Scale
Brief Title: Correlation Between Quality of Life and Severity of Parkinson's Disease
Status: Completed | Type: Observational
Sponsor: R.O.M.A. - Rehabilitation & Outcome Measures Assessment (Other)
Responsible Party: Principal Investigator, Giovanni Galeoto, Department of Public Health and Infection disease, Sapienza University of Rome, R.O.M.A. - Rehabilitation & Outcome Measures Assessment
Other Study IDs: Quality of Life and Parkinson
Record Dates: First submitted 2019-09-28; First posted 2019-10-01 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Parkinson Disease; Quality of Life
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — All participants were evaluated with the PDQ-39, and the severity of PD was recorded according to the H&Y scale by a neurologist.

SUMMARY:
This study aim to evaluate the correlation between Quality of Life (QoL) and severity of Parkinson's Disease (PD) by assessing the presence of an optimal cut-off point on the Parkinson's disease questionnaire (PDQ-39) as related to the Hoehn & Yahr (H&Y) scale in a cohort of Italian adults with PD.

A multicenter, cross-sectional study was performed in central and northern Italy. This study was conducted on a cohort of consecutive individuals at three neurologic outpatient clinics. All participants were evaluated with the PDQ-39, and the severity of PD was recorded according to the H&Y scale by a neurologist. Receiver operating characteristic (ROC) curves and coordinates of the curve, which were visually inspected, were used to find cut-off points with optimal sensitivity and specificity. These were in turn used to determine the optimal PDQ-39 cut-off score for identifying disease severity according to H&Y stages.

ELIGIBILITY:
Inclusion Criteria:

* age > 50 but < 90 years,
* H&Y stages I, II, III, and IV,
* a mini-mental state examination > 22 points,
* a minimum level of five years of education.

Exclusion Criteria:

* Individuals with emotional or psychiatric problems (as determined by clinical screening)

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Fivehundred thirteen individuals with Parkinson's Disease (PD) were recruited, all of whom agreed to participate and were thus included in the study. From the general analysis resulted that the greatest number of participants were stage II, according to Hoehn & Yahr (H&Y), followed by stage III, stage I, and finally stage IV. Participants between the age of 50 and 69 were mainly stage I or II, while participants aged 70 to 89 had a greater severity of PD (stage II and III). Most women were in H&Y stage II and III, while most men were mainly in stage II, followed by stage I and III, with a very similar number of participants. A common result for all analyses was the presence of a very low number of participants with stage IV.
Sampling Method: Non-Probability Sample
Enrollment: 513 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-03-25 (Actual); Study Completion 2019-09-25 (Actual)

PRIMARY OUTCOMES:
Hoehn & Yahr (H&Y) | at admission to the neurologic outpatient clinics
  severity of Parkinson's disease
Parkinson's Disease questionnaire (PDQ-39) | at admission to the neurologic outpatient clinics
  quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Human Neurosciences, Sapienza University of Rome, Roma, RM, Italy

IPD SHARING:
Plan to Share IPD: Yes